CLINICAL TRIAL: NCT06817733
Title: Clinical Study on Prostate Thermal Vapor Ablation Guided by MRI/TRUS Fusion Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qing Yuan, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REZUM2025
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign prostatic hyperplasia; Rezum; MRI-TRUS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Rezum (Experimental): Participants in this group will undergo transurethral thermal vaporization of the prostate.
  Interventions: Procedure: Transurethral Thermal Vaporization of the Prostate

INTERVENTIONS:
Procedure: Transurethral Thermal Vaporization of the Prostate — After anesthesia, the patient is placed in the lithotomy position, and standard aseptic preparation and draping are performed. A cystoscope and a transrectal ultrasound (TRUS) probe are inserted. Following real-time image fusion and localization according to the preoperative plan, needles are inserted to deliver thermal vaporization to the prostate. Each needle treatment lasts 8 seconds, and the entire procedure is completed within 200 seconds after activation of the needle pathway.

SUMMARY:
Objective of the Clinical Trial

The objective of this clinical trial is to preliminarily assess the feasibility and safety of performing precise prostate thermal vapor ablation under MRI/TURS guidance. The primary questions it aims to address are:

Can precise prostate thermal vapor ablation under MRI/TURS guidance effectively treat benign prostatic hyperplasia (BPH) and alleviate lower urinary tract symptoms (LUTS)? What safety issues may arise in participants after undergoing prostate thermal vapor ablation? Study Procedures Participants Preoperative Evaluation: Participants will undergo comprehensive preoperative assessments, including clinical examinations and laboratory tests.

Procedure: Participants will receive precise prostate thermal vapor ablation under MRI/TURS guidance.

Postoperative Follow-up:

Regular follow-up to reassess prostate volume. Periodic completion of the International Prostate Symptom Score (IPSS) questionnaire.

Regular measurement of maximum urinary flow rate (Qmax) and post-void residual urine volume (PVR).

Research Team The research team will conduct precise prostate thermal vapor ablation under MRI/TURS guidance for the participants and manage their follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-85 years;
* International Prostate Symptom Score (IPSS) ≥ 8, indicating moderate to severe Lower Urinary Tract Symptoms (LUTS) that significantly impact quality of life;
* Poor response to pharmacological treatment or refusal of pharmacological treatment;
* Prostate volume 30-80 mL;
* Maximum urinary flow rate (Qmax) < 15 mL/s;
* Post-void residual urine volume (PVR) < 300 mL;
* Willingness to provide informed consent and participate in postoperative follow-up.

Exclusion Criteria:

* Prostate volume < 30 mL or > 80 mL;
* Severe urinary tract infection;
* Preoperative definitive diagnosis of prostate cancer;
* Known neurogenic bladder, detrusor muscle weakness, urethral stricture, or other non-BPH causes of urinary obstruction;
* Patients with prostatitis;
* History of invasive prostate interventions, such as radiofrequency ablation, laser therapy, or microwave treatment;
* Patients with severe cardiovascular disease, chronic obstructive pulmonary disease, severe diabetes, hepatic or renal dysfunction, or systemic bleeding disorders, as assessed by the investigator to be unsuitable for surgery.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume changes in the prostate transition zone | From enrollment to 6 months after surgery
  The volume of the transitional zone measured by MRI before and 6 months after surgery

SECONDARY OUTCOMES:
Prostatic volume change | From enrollment to 6 months after surgery
  Changes in prostate volume before and 6 months after surgery
IPSS | From enrollment to 6 months after surgery
  International Prostate Symptom Score.The minimum IPSS score was 0, the maximum was 35, and the higher the score, the more severe the lower urinary tract symptoms were. 0-7 was classified as mild symptoms, 8-19 as moderate symptoms, and 20-35 as severe symptoms.
Qmax | From enrollment to 6 months after surgery
  Maximum urine flow rate
PVR | From enrollment to 6 months after surgery
  Post-Void Residual urine
Duration of postoperative indwelling urinary catheter | From the end of the procedure until the catheter is removed.It is estimated that the longest time will not exceed 2 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doppalapudi SK, Gupta N. What Is New with Rezum Water Vapor Thermal Therapy for LUTS/BPH? Curr Urol Rep. 2021 Jan 6;22(1):4. doi: 10.1007/s11934-020-01018-6. PMID 33403529
- [Result] Ines M, Babar M, Singh S, Iqbal N, Ciatto M. Real-world evidence with The Rezum System: A retrospective study and comparative analysis on the efficacy and safety of 12 month outcomes across a broad range of prostate volumes. Prostate. 2021 Sep;81(13):956-970. doi: 10.1002/pros.24191. Epub 2021 Jul 12. PMID 34254333
- [Result] McVary KT, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Pliskin M, Beahrs JR, Prall D, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Tadros NN, Gange SN, Roehrborn CG. Final 5-Year Outcomes of the Multicenter Randomized Sham-Controlled Trial of a Water Vapor Thermal Therapy for Treatment of Moderate to Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2021 Sep;206(3):715-724. doi: 10.1097/JU.0000000000001778. Epub 2021 Apr 19. PMID 33872051
- [Result] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Result] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Result] Sandhu JS, Bixler BR, Dahm P, Goueli R, Kirkby E, Stoffel JT, Wilt TJ. Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia (BPH): AUA Guideline Amendment 2023. J Urol. 2024 Jan;211(1):11-19. doi: 10.1097/JU.0000000000003698. Epub 2023 Sep 14. PMID 37706750
- [Result] Zhang W, Zhang X, Li H, Wu F, Wang H, Zhao M, Hu H, Xu K. Prevalence of lower urinary tract symptoms suggestive of benign prostatic hyperplasia (LUTS/BPH) in China: results from the China Health and Retirement Longitudinal Study. BMJ Open. 2019 Jun 19;9(6):e022792. doi: 10.1136/bmjopen-2018-022792. PMID 31221864
- [Result] Lee SWH, Chan EMC, Lai YK. The global burden of lower urinary tract symptoms suggestive of benign prostatic hyperplasia: A systematic review and meta-analysis. Sci Rep. 2017 Aug 11;7(1):7984. doi: 10.1038/s41598-017-06628-8. PMID 28801563